CLINICAL TRIAL: NCT05162079
Title: Protocol for the ESREFLUJO Study: Epidemiological Study of Heartburn and Gastroesophageal Reflux in Community Pharmacy
Acronym: ES-REFLUJO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Elsa López Pintor, Lecturer, Universidad Miguel Hernandez de Elche
Other Study IDs: SEFAC1.20I.
Record Dates: First submitted 2021-11-16; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Reflux
Keywords: HEARTBURN, DYSPEPSIA, REFLUX, PHARMACY
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Symptoms as heartburn and/or reflux is frequent consultations in community pharmacies, the characterization of them is crucial to provide appropriate patient counseling. To facilitate the assistance work of the community pharmacist and its coordination between different levels of care, a group of experts in Community Pharmacy, Primary Care, and Gastroenterology has recently worked on an algorithm to manage these symptoms.

Objective: Analyse the epidemiological characteristics of patients who consult for symptoms of heartburn and/or reflux in Spanish community pharmacies, and evaluate the clinical and humanistic results of the protocolization of a Professional Pharmaceutical Service in said patients.

Methods and analysis: The study design consists of a cross-sectional descriptive part, in which the clinical and sociodemographic characteristics of the patients who come to the community pharmacy will be evaluated for consultation derived from heartburn and/or reflux symptoms and a before-after descriptive study in which will evaluate the clinical and humanistic results in patients who come to the pharmacy after receiving pharmaceutical care.

ELIGIBILITY:
Inclusion Criteria:

* Population´s age ≥ 18 years
* Patients who consult for mild symptoms of heartburn and/or gastroesophageal reflux or request treatment for it.

Exclusion Criteria:

* Subjects who request treatment for symptoms of heartburn and/or gastroesophageal reflux for another person
* Women with high-risk pregnancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Spanish patients who visit the pharmacies asking for advice of acid-reflux symptoms or requesting non-prescription medication for it
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Collection of sociodemographic data of participants | 8 minutes each questionnaire
  At the initial visit, sociodemographic variables will be collected through a Data Collection Notebook (CDR): sex, age, level of education, employment status, civil status.
Collection of clinical data of participants | 8 minutes each questionnaire
  At the initial visit, clinical data will be collected through a Data Collection Notebook (CDR):
  * Risk factors: Body mass index (BMI), smoking, food consumption
    • Weight and height will be combined to report BMI in kg/m^2.
  * Symptoms throught the questionnaire: The Gastro-oesophageal Reflux Disease Impact Scale (GIS)
  * Treatments or medications used
Detail the evolution of the patient's symptoms 14 days after intervention | 5 minutes
  An independent external monitor will make a telephone call to each patient to collect the evolution of the patient´s symptoms through a questionnaire: The Gastro-oesophageal Reflux Disease Impact Scale (GIS). It is a scale of frequency, the lower scores mean better health in the patient less frequency of disturbances)
Evaluate patient satisfaction | 5 minutes
  An independent external monitor will make a telephone call to each patient to collect the evolution of the patient´s symptoms through a questionnaire: Degree of satisfaction with the pharmaceutical care received (The score is the level of agreement, high punctuation means more satisfaction) and If the patient gets medication: Treatment Satisfaction Questionnaire for Medication (TSMQ, v1.4). (The score is the level of satisfaction, high punctuation means more satisfaction)

REFERENCES:
- [Derived] Puig-Molto M, Lumbreras B, Lopez-Pintor E. Improving Proton-Pump Inhibitor Adherence Intervention Between Primary Care and Community Pharmacies: A Pre-Post Intervention Study. Patient Prefer Adherence. 2024 Dec 18;18:2569-2580. doi: 10.2147/PPA.S485307. eCollection 2024. PMID 39713795
- [Derived] Lopez-Pintor E, Puig-Molto M, Lumbreras B. EsReflux Protocol: Epidemiological Study of Heartburn and Reflux-like Symptoms in Spanish Community Pharmacies. Int J Environ Res Public Health. 2022 Aug 9;19(16):9807. doi: 10.3390/ijerph19169807. PMID 36011453